CLINICAL TRIAL: NCT04127942
Title: Six-month Efficacy of Ultrasound-guided Platelet-rich Plasma Injection for Temporomandibular Disorders
Brief Title: Platelet-rich Plasma Injection for Temporomandibular Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no sufficient enrolled pateints
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Clinical Professor of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-106-05-026
Record Dates: First submitted 2019-04-22; First posted 2019-10-16 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Temporomandibular Disorder
Keywords: platelet-rich plasma; ultrasound guided injection.; Temporomandibular disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: access the efficacy of ultrasound-guided PRP injection therapy of TMD, with normal saline used as control group.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet-rich plasma injection (Experimental): 1cc platelet-rich plasma(PRP) injection in the superior temporomandibular disk joint space by ultrasound guidance.
  Interventions: Procedure: platelet-rich plasma injection therapy of TMD
- normal saline injection (Placebo Comparator): 1cc normal saline injection in the superior temporomandibular disk joint space by ultrasound guidance.
  Interventions: Procedure: platelet-rich plasma injection therapy of TMD

INTERVENTIONS:
Procedure: platelet-rich plasma injection therapy of TMD — The administer injected 1cc PRP in the superior temporomandibular disk joint space by ultrasound guidance.

SUMMARY:
Temporomandibular disorder (TMD) involves the temporomandibular joint (TMJ) and surrounding structure, causing problems including myofascial pain and joint degeneration. TMD is mostly seen in the age group of 18 to 44. TMD treatment includes conservative (non-surgical) and surgical treatment. Surgical TMD treatment has a decent success rate but requires general anesthesia, hospital stay and surgical incision. There are also some risks of facial nerve and vascular damage, infection, puncture to middle cranial fossa. Conservative treatments include medication , physical therapy, use of occlusal splint, hyaluronic acid (HA) or Botulinum toxin injection and concentrated glucose solution. However, those managements lack the evidence from large placebo-controlled clinical trials. Therefore, the development of novel non-surgical treatment is important and of great potential. The ultrasound guidance provides visualization of the lesion site, allowing the operator to provide injection precisely and avoid damage on adjacent tissue, nerves and vessels. it is not only convenient and economic, but also associated with significantly less radiation exposure than conventional techniques such as computer tomography or fluoroscopy. Using ultrasound guidance in injective TMD treatment can increase successful rate and prevent unnecessary side effects. While current available evidences suggest the promising effect of platelet-rich plasma (PRP) injection therapy in treating TMD, publication of study with strict design is still lacking. Therefore, this study is a randomized, controlled and double-blind design, which aimed to access the efficacy of ultrasound-guided PRP injection therapy of TMD, with normal saline used as control. Looking forward to establish TMD clinical treatment guideline in the future.

DETAILED DESCRIPTION:
Objectives:

Temporomandibular disorder (TMD) involves the temporomandibular joint (TMJ) and surrounding structure, causing problems including myofascial pain and joint degeneration. TMD is mostly seen in the age group of 18 to 44. TMD treatment includes conservative (non-surgical) and surgical treatment. Surgical TMD treatment has a decent success rate but requires general anesthesia, hospital stay and surgical incision. There are also some risks of facial nerve and vascular damage, infection, puncture to middle cranial fossa. Conservative treatments include medication , physical therapy, use of occlusal splint, hyaluronic acid (HA) or Botulinum toxin injection and concentrated glucose solution. However, those managements lack the evidence from large placebo-controlled clinical trials. Therefore, the development of novel non-surgical treatment is important and of great potential. The ultrasound guidance provides visualization of the lesion site, allowing the operator to provide injection precisely and avoid damage on adjacent tissue, nerves and vessels. it is not only convenient and economic, but also associated with significantly less radiation exposure than conventional techniques such as computer tomography or fluoroscopy. Using ultrasound guidance in injective TMD treatment can increase successful rate and prevent unnecessary side effects. While current available evidences suggest the promising effect of platelet-rich plasma (PRP) injection therapy in treating TMD, publication of study with strict design is still lacking. Therefore, this study is a randomized, controlled and double-blind design, which aimed to access the efficacy of ultrasound-guided PRP injection therapy of TMD, with normal saline used as control. Looking forward to establish TMD clinical treatment guideline in the future.

Methods:

The out-patients with unilateral or bilateral TMD、joint mobility dysfunction or joint noise from this hospital were enrolled. They were randomized via computer into 2 groups (PRP group and normal saline group). There are 30 patients in each group. The PRP group received 1cc PRP injection in the superior temporomandibular disk joint space by ultrasound guidance. The normal saline group received the same procedure as PRP group with 1 cc normal saline injection. Both group received the same protocol of physical therapy (manual therapy, stretching exercise, posture training with 30 minutes per session and 2 sessions per weeks) for 12 weeks. Those physical therapies were under the guidance of one therapist who didn't know the patient's allocation.

The investigator and subjects did not know the group assignment. Evaluations were performed at time points prior to injection and 2 weeks, 1st, 3rd , and 6th months post injection by one doctor (who didn't know about the group assignment). Evaluations include Visual Analogue Scale (VAS) of the degree of pain, masticatory efficiency, perceived joint noise and measure of maximal interincisal opening, painless oral opening, mandibular lateral movement and protrusion movement. The investigator also evaluated symptoms or signs of side effects and complications.

Besides, the subjects can't receive any treatment include medications or injection for pain control, but allowed to take Acetaminophen 500mg, maximal dosage 4g per day to relieve refractory pain during follow up period. If any participant broke the rules or took Acetaminophen over daily dosage, the participant will be excluded to this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Duration of symptoms ( temporomandibular joint pain or tenderness, joint noise or joint motility dysfunction)more than 3 months.
* Diagnosis was confirmed by using the original Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) and the severity at least Grade II.

Exclusion Criteria:

* Head and neck cancer
* Neurological disease
* Cognition impairment
* Coagulopathy
* Pregnancy
* Inflammation status
* Infection status
* Previously undergone wrist surgery or steroid injection for TMD

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of the degree of pain | 6 months
  *. Visual Analogue Scale of the degree of pain: with the score ranging from 10 (tremendous pain) to 0 (no pain).

SECONDARY OUTCOMES:
measure of maximal interincisal opening and painless mouth opening | 6 months
  The subject was instructed, "Open your mouth as wide as possible without causing pain or discomfort." Then, using ruler to measured the intercisal distance (cm) by placing the ruler between central incisors.
measure of maximal mandibular excursion and protrusion. | 6 months
  * Excursion: Vertical marks were made on the anterior surface of the lower central incisors in relationship to the upper central incisors and the subject was instructed to "move your jaw as far to the side as you can comfortably." The measurement was taken as the horizontal distance between the 2 marks when the jaw was moved to the left and the right by using ruler to measured the intercisal distance (cm)
  * Protrusion: Two vertical lines were made on the first upper and lower canine incisors. The subject was instructed to "move your jaw as far forward as you can." The measurement was taken as the distance between the 2 marks by using ruler to measured the intercisal distance (cm)
Visual Analogue Scale of masticatory efficiency | 6 months
  *. Visual Analogue Scale of masticatory efficiency:with the score ranging from 10 (good; can eat solid food) to 0 (poor; only liquid diet)
Visual Analogue Scale of perceived joint noise | 6 months
  *. Visual Analogue Scale of perceived joint noise: with the score ranging from 10 (much noise) to 0 (no noise).

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD,MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper BC, Kleinberg I. Examination of a large patient population for the presence of symptoms and signs of temporomandibular disorders. Cranio. 2007 Apr;25(2):114-26. doi: 10.1179/crn.2007.018. PMID 17508632
- [Background] Gencer ZK, Ozkiris M, Okur A, Korkmaz M, Saydam L. A comparative study on the impact of intra-articular injections of hyaluronic acid, tenoxicam and betametazon on the relief of temporomandibular joint disorder complaints. J Craniomaxillofac Surg. 2014 Oct;42(7):1117-21. doi: 10.1016/j.jcms.2014.01.041. Epub 2014 Feb 4. PMID 24853591
- [Background] Martins WR, Blasczyk JC, Aparecida Furlan de Oliveira M, Lagoa Goncalves KF, Bonini-Rocha AC, Dugailly PM, de Oliveira RJ. Efficacy of musculoskeletal manual approach in the treatment of temporomandibular joint disorder: A systematic review with meta-analysis. Man Ther. 2016 Feb;21:10-7. doi: 10.1016/j.math.2015.06.009. Epub 2015 Jun 25. PMID 26144684
- [Background] Kummoona R. Surgical managements of subluxation and dislocation of the temporomandibular joint: clinical and experimental studies. J Craniofac Surg. 2010 Nov;21(6):1692-7. doi: 10.1097/SCS.0b013e3181f3c682. PMID 21119402
- [Background] Sivri MB, Ozkan Y, Pekiner FN, Gocmen G. Comparison of ultrasound-guided and conventional arthrocentesis of the temporomandibular joint. Br J Oral Maxillofac Surg. 2016 Jul;54(6):677-81. doi: 10.1016/j.bjoms.2016.04.004. Epub 2016 Apr 23. PMID 27118616
- [Background] Fernandez-Ferro M, Fernandez-Sanroman J, Blanco-Carrion A, Costas-Lopez A, Lopez-Betancourt A, Arenaz-Bua J, Stavaru Marinescu B. Comparison of intra-articular injection of plasma rich in growth factors versus hyaluronic acid following arthroscopy in the treatment of temporomandibular dysfunction: A randomised prospective study. J Craniomaxillofac Surg. 2017 Apr;45(4):449-454. doi: 10.1016/j.jcms.2017.01.010. Epub 2017 Jan 25. PMID 28237253